CLINICAL TRIAL: NCT02907723
Title: Assessment of a Wrist Device Recording Sleep Parameters, Before and After Deep Brain Stimulation for Parkinson's Disease
Brief Title: Feasibility of Continuous Sleep Recording in Patients Undergoing Deep Brain Stimulation for Parkinson's Disease
Acronym: BRACELET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JBL_2014_11
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Polysomnography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous Sleep Recording (Experimental): Continuous Sleep Recording in Patients
  Interventions: Device: Sleep Recording

INTERVENTIONS:
Device: Sleep Recording — the device records movements during patients' sleep

SUMMARY:
This pilot study aims to assess a new device designed for an objective measure of sleep parameters. The purpose of the device is to assess, in a more simple and precise way, the impact of deep brain stimulation on patient's sleep.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18 years old
* with Parkinson disease
* scheduled for implantation of electrodes for deep brain stimulation

Exclusion criteria:

* pregnant or breast feeding patient
* refusal to participate in the study
* patient under legal protection
* no health insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
mean sleep duration per night | 15 days
mean sleep onset latency | 15 days
mean number of awakenings per night | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe BRANDEL, MD, Principal Investigator — Fondation OPH A de Rothschild